CLINICAL TRIAL: NCT04077359
Title: Prospective Trial for Examining Hematuria Using Computed Tomography
Acronym: PROTEHCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Responsible Party: Principal Investigator, Erik Rud, Consulting radiologist, PhD, Oslo University Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2019/395
Record Dates: First submitted 2019-08-30; First posted 2019-09-04 (Actual); Last update posted 2022-09-06 (Actual); Status verified 2022-09

CONDITIONS: Urothelial Carcinoma; Renal Cell Carcinoma; Renal Cyst; Renal Stone
MeSH Terms: conditions — Carcinoma, Transitional Cell; Carcinoma, Renal Cell; Nephrolithiasis

STUDY DESIGN:
Intervention Model Description: One sample, paired, non-inferiority study with a 7.5% non-inferiority limit. Each patient undergo the experimental CT and the control CT
Masking Description: one investigator evaluates the experimental arm a second investigator evaluates the control arm without knowledge of the other
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- nephrographic phase CT (Experimental): the nephrographic phase will be evaluated alone by a radiologist blinded to the remaining series
  Interventions: Diagnostic Test: CT
- gold standard (Active Comparator): all series (unenhanced, corticomedullary, nephrographic and excretory phase) will be evaluated by a radiologist not involved in the experimental arm
  Interventions: Diagnostic Test: CT

INTERVENTIONS:
Diagnostic Test: CT — the CT consist of four phases; non-enhanced, corticomedullary, nephrographic and excretory phase.

SUMMARY:
The primary objective is to evaluate whether one-phase nephrographic CT (experimental) is sufficient to detect urothelial cell carcinoma in patients with hematuria compared to the traditional four-phase CT (control).

DETAILED DESCRIPTION:
Responsible centers Oslo University Hospital, Aker. Division of Radiology and Nuclear medicine.

Study type: Prospective clinical trial

Study design: One sample paired proportion, non-inferiority study with a 7.5% non-inferiority limit.

Investigational product: One phase nephrographic CT (experimental arm) vs. Four-phase CT (control arm)

Objective:The primary objective is to evaluate whether one-phase nephrographic CT (experimental) is sufficient to detect urothelial cell carcinoma in patients with asymptomatic macroscopic hematuria compared to the traditional four-phase CT (control).

Primary endpoints: The difference in accuracy between the experimental- and control arm.

there will also be a secondary reading in order to asses interobserver variability for both the experimental and the control arm

Sample size: 250 patients

ELIGIBILITY:
Inclusion Criteria:

* Asymptomatic macroscopic hematuria referred to CTU before cystoscopy
* >18 years old

Exclusion Criteria:

* Symptomatic urinary tract infection relieved by antibiotics
* Patients referred to CTU after cystoscopy
* Cystoscopy within the last 6 months
* Symptomatic stone disease
* Macroscopic hematuria after recent catherization or instrumentation
* Microscopic hematuria
* Previous history of Urothelial cell carcinoma
* Known staghorn calculi
* Allergy to iodine contrast media
* Impaired renal function (eGFR < 30m/min/1.73m2)
* Unable to provide consent for any reason
* For any reason, do not wish to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2019-09-15 (Actual); Primary Completion 2021-07-01 (Actual); Study Completion 2021-07-01 (Actual)

PRIMARY OUTCOMES:
accuracy for detecting urothelial cell carcinomas | all examinations are evaluated immediately after the CT examination. Follow-up ascertainment of UCC diagnosis after one year
  the accuracy of the experimental arm will not be worse than the accuracy of the control CT by a margin of more than 7.5%

SECONDARY OUTCOMES:
false negative rate | all examinations are evaluated immediately after the CT examination
  The difference in false negative rates
false positive rate | all examinations are evaluated immediately after the CT examination
  The difference in false positive rates
renal cell carcinoma detection rates | all examinations are evaluated immediately after the CT examination. Follow-up ascertainment of RCC diagnosis after one year
  The detection rates in the two arms
Area under the curve (AUC) | all examinations are evaluated immediately after the CT examination
  the difference in AUC of the two arms
predictive values | all examinations are evaluated immediately after the CT examination
  The difference in the predictive values of the two arms
Detection or urinary calculi | all examinations are evaluated immediately after the CT examination
  The difference in detection of the two arms
Detection of Bosniak cyst | all examinations are evaluated immediately after the CT examination
  The difference in detection in the two arms
Interobserver variability | all examinations are evaluated immediately after the CT examination
  The agreement and variability between primary and secondary readers

CONTACTS AND LOCATIONS:
Overall Officials: Erik Rud, Principal Investigator — Oslo University Hospital
Locations (1):
- Oslo University Hospital, Oslo, Norway